CLINICAL TRIAL: NCT03937895
Title: Phase 1/2a Clinical Trial for the Evaluation of Safety and Efficacy of Allogeneic NK Cell ("SMT-NK") in Combination With Pembrolizumab for Patients With Gemcitabine-refractory Biliary Tract Cancer
Brief Title: Allogeneic NK Cell ("SMT-NK") in Combination With Pembrolizumab in Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SMT bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNK-SIT-02
Record Dates: First submitted 2019-04-29; First posted 2019-05-06 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Biliary Tract Cancer
Keywords: Biliary Tract Cancer; BTC; Cholangiocarcinoma
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: single arm (Experimental): * Biological: 'SMT-NK' Inj. (allogeneic Natural Killer cell) weekly administration for 2 weeks. After that, 1 week is a withdrawal period. (Phase 1: up to *cycle 3, Phase 2a: up to cycle 9)
  * Drug: Pembrolizumab administration of Pembrolizumab 200mg/m2 at first week during cycle.
    * Cycle: 1 cycle is 3 weeks in total.'SMT-NK' Inj is administered at first and second week, and Pembrolizumab is administered at first week. The third week is a withdrawal period.
  Interventions: Biological: 'SMT-NK' Inj (allogeneic Natural Killer cell); Drug: Pembrolizumab Injection [Keytruda]

INTERVENTIONS:
Biological: 'SMT-NK' Inj (allogeneic Natural Killer cell) — In 120 mL, 3x10^6 (± 20%) cells/kg. weekly administration via Intravenous for 2 weeks. After that, 1 week is a withdrawal period.
Drug: Pembrolizumab Injection [Keytruda] — Administration via Intravenous of 200 mg every 3 weeks(one administration per cycle.).

SUMMARY:
The term of biliary tract cancer (BTC) or cholangiocarcinoma refers to all tumors that arise from the biliary tract or the biliary drainage system, including the gallbladder. According to the data from National Cancer Information Center in 2016, annual incidence of the cancer in Korea is 6,685 (13.1 per 100,000 population) which corresponds to about 2.9% of all cancers.

BTC is one of the most prognostic cancer with less than 30% of 5-year survival rate and the case with long-term survival can be possibly done with early detection of the cancer. However, most of BTC is found in advanced stages due to the difficulty of early detection, resulting in that the 5-year survival rate of the advanced BTC becomes less than 3%. More than 50% of the patients depends on Gemcitabine based chemotherapy but response rate of the chemotherapy remains around 30%. Thus, improving the survival rate with the standard chemotherapy is very limited and furthermore selection of second-line therapy is not easy. For this reason, development of an alternative therapeutic agent is urgently required.

NK (natural killer) cells are important cytotoxic innate immune cells that are involved in the elimination of cancer cells. Two main NK cell subsets have been defined on the basis of CD56 and CD16 expression: CD56^brightCD16- NK subset produces abundant cytokines including interferon-γ (IFN-γ) and tumor necrosis factor-α, whereas CD56^dimCD16+ NK subpopulation has high cytolytic activity and releases the granules containing perforin and granzymes.

Various clinical studies have been conducted to treat cancers using NK cells worldwide including Korea and therapeutic clinical results are shown for various cancers. The clinical application of NK cells is carried out by culturing and activating the NK cells isolated from blood of either patient (autologous) or blood donor (allogeneic). Recently, NK cell therapy for cholangiocarcinoma has been successfully done (NCT03358849) with allogeneic NK cell, showing safety and potential efficacy.

Like T cells, a recent study with digestive cancer has shown that NK cells also express PD-1, especially with more number of PD-1 in cancer patients than in healthy individuals, suggesting that blocking PD-1 can be used as a potential strategy to increase the anticancer activity of NK cells. Therefore, combined therapy with the immune-check point such as pembrolizumab can be useful in elevating the anticancer activity of NK cells.

ELIGIBILITY:
[Inclusion Criteria]

Patients who received a histopathological or cytologic diagnosis of nonresectable, advanced biliary tract carcinoma (intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer) and patients with refractory disease after chemotherapy and/or patients who have difficulty with chemotherapy due to side effects of chemotherapy.

1. A person who receives an explanation from the trial manager about the purpose, contents, and characteristics of the Investigational products for the clinical trial and is signed by the person, guardian or legal representative in the written informed consent.
2. Be ≥19 years of age on day of signing informed consent.
3. Histopathological or cytologic diagnosis of advanced adenocarcinoma of the biliary tract.
4. Have a performance status of ≤2 on the ECOG Performance Scale.
5. Patients who survival period is expected to be at least 3 months.
6. Patients who meet the following conditions:

   * ANC(Absolute Neutrophil Count) ≥ 1,500/μL
   * Hemoglobin≥ 10 g/dL
   * Platelet> 100,000/μL
   * Serum BUN & Creatinine ≤ 1.5 x upper limit of normal (ULN)
   * AST & ALT ≤ 2.5 x upper limit of normal (ULN)
   * Bilirubin ≤ 3mg/L
7. Patients who agreed to the allogeneic natural killer cells therapy separated from the family of the patient or healthy donor's blood.
8. Patients have a negative serum or urine pregnancy test (HCG, human chorionic gonadotropin) within 72 hours prior to receiving the first dose of study medication and agreed to use 2 methods of contraception. The period of contraception is up to 6 months after the last administration of Pembrolizumab.
9. Patients who meet one or more of the following conditions.

   * Patients have at least 1% Combined Positive Score (*CPS) PD-L1 expression detected on the tumor, as determined by **immunohistochemistry performed by a central laboratory.

     *CPS = (number of PD-L1 positive tumor cells, lymphocytes, macrophage)/ (total number of viable tumor cells) X 100

     **immunohistochemistry: IHC 22C3 pharmDx test
   * Patients who have a positive *MSI-H or **dMMR test.

     * MSI-high positive tumors analyzed by PCR.
     * dMMR positive tumors analyzed by immunohistochemical staining .

       * *MSI-H was measured by PCR, and positive finding when two or more unstable markers were detected in PCR for 5 microsatellite markers.
       * **dMMR is analyzed by immunohistochemical staining and positive when the discovery of one or more genes in MLH1, MSH2, MSH6 and PMS2 staining is lost.

[Exclusion Criteria]

1. Patients who have previous history of Immune deficiency or autoimmune disease that can be aggravated by immunotherapy(for example: Rheumatoid arthritis, systemic lupus erythematosus, vasculitis, multiple sclerosis, Crohn's disease, ulcerative colitis, adolescent-developed insulin-dependent diabetes mellitus).
2. Diagnosis of immunodeficiency or is receiving systemic steroid therapy.
3. Have with pneumonia, colitis, hepatitis, nephritis, endocrine disorders(for example: Pituitary gland, thyroid dysfunction, Type 1 diabetes, etc.) associated with immunodeficiency.
4. Other malignant tumors within 5 years before the study enrollment.
5. Previous history of anti-angiogenic agent treatment before the study enrollment.
6. Received chemotherapy not less than 4 weeks old before the first administration of investigational products.
7. Apparent myocardial infarction or uncontrolled arterial hypertension.
8. Serious allergic history.
9. Serious mental illness.
10. Female who are pregnant, breastfeeding or intending to become pregnant during the study period.
11. A person who participated in another clinical trial within 4 weeks prior to the start of the study(based on the date of signing the informed consent.).
12. Previously administrated Pembrolizumab and other anti-PD-1/PD-L1 agent.
13. Previously administrated natural killer cell.
14. Patients who did not resolve the adverse event of the drug administered 4 weeks prior to enrollment.
15. Previous history of active central nervous system (CNS) metastasis and/or carcinomatous meningitis.
16. Previous history of non-infectious pneumonia.
17. Previous history of Has an active infection requiring systemic therapy.
18. Previous historyof Human Immunodeficiency Virus (HIV).
19. Previous history of active Hepatitis B (e.g., HBsAg reactive), Hepatitis C, Active tuberculosis.
20. Have received a live vaccine within 4 weeks before the first administration of investigational products.
21. Hypersensitivity to Pembrolizumab additive.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Phase 1 - Dose Limiting Toxicity of the dose of 'SMT-NK' Inj. in combination with Pembrolizumab. | Up to 9 weeks from Baseline.
  DLT (Dose Limiting Toxicity) Assessment
Phase 2a - Objective Response Rate (ORR) | Up to 27 weeks from Baseline.
  ORR (Objective Response Rate, sum of PR and CR) is finally evaluated In the third tumor response evaluation by CT(according to RECIST V1.1).

SECONDARY OUTCOMES:
Phase 2a - Time to Progression | Up to 39 weeks from Baseline
  The length of time from the baseline until determine to progressive disease(PD).
Phase 2a - Toxicity (according to CTCAE 5.0) | Up to 39 weeks from Baseline
  Levels of adverse events and changes of experimental parameters are described according to CTCAE (version 5.0). Defined as incidence and severity of adverse events, significant laboratory changes, changes in vital signs, incidence of concomitant medications, changes from baseline over time in ECOG PS/100-mm Visual Analog Score for pain, incidence of dose adjustments over the treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Seung Woo Park, MD. PhD, Principal Investigator — Division of Gastroenterology, Department of Internal Medicine, Yonsei University College of Medicine, Severance Hospital
Locations (2):
- South Korea (2):
  - Severance Hospital, Seoul
  - Gangnam Severance Hospital, Seoul

REFERENCES:
- See also: Phase 1 Clinical Trial to Evaluate the Safety of Allogeneic NK Cell ("SMT-NK") Cell Therapy in Advanced Biliary Tract Cancer — https://clinicaltrials.gov/ct2/show/study/NCT03358849?term=Nk+cell&cond=biliary+tract+cancer&cntry=KR&rank=1